CLINICAL TRIAL: NCT06150573
Title: A Randomized, Controlled, Single-Blind Clinical Study Assessing the Effects of an Experimental Dentifrice in Maintaining Tooth Color Following Tooth Bleaching
Brief Title: A Study Assessing the Effects of an Experimental Dentifrice in Maintaining Tooth Color Following Tooth Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300109
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Dentin Sensitivity; Oral Hygiene
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Dentifrice (Experimental): Participants will dose the toothbrush provided with a strip of test dentifrice (5% KNO3, 1% alumina, 5% STP and 1150 parts per million [ppm] fluoride as sodium fluoride) and will brush for two timed minutes twice daily (morning and evening) for up to 27 weeks (dentifrice will be used for 2 weeks pre peroxide, 1 week during peroxide and 24 weeks post peroxide application). At Week 3, participants will perform the first application of peroxide tooth bleaching as per the instructions provided and continue the application daily for up to 7 days.
  Interventions: Drug: Test Dentifrice
- Reference Dentifrice (Active Comparator): Participants will dose the toothbrush provided with a strip of reference dentifrice (dentifrice containing 1150 ppm fluoride as sodium fluoride) and will brush for two timed minutes twice daily (morning and evening) for up to 27 weeks (dentifrice will be used for 2 weeks pre peroxide, 1 week during peroxide and 24 weeks post peroxide application). At Week 3, participants will perform the first application of peroxide tooth bleaching as per the instructions provided and continue the application daily for up to 7 days.
  Interventions: Drug: Reference Dentifrice (Aquafresh Cavity Protection)

INTERVENTIONS:
Drug: Test Dentifrice — Dentifrice containing 5% weight by weight (w/w) KNO3, 1% alumina, 5% STP and 1150 ppm fluoride as sodium fluoride.
  Arms: Test Dentifrice
Drug: Reference Dentifrice (Aquafresh Cavity Protection) — Dentifrice containing 1150 ppm fluoride as sodium fluoride.
  Arms: Reference Dentifrice

SUMMARY:
The main aim of this study is to investigate the ability of an experimental dentifrice containing 5 percent (%) potassium nitrate (KNO3), 1% alumina and 5% sodium tripolyphosphate (STP), to maintain tooth color and reduce extrinsic dental stain accumulation following peroxide tooth bleaching compared to a regular fluoride dentifrice.

DETAILED DESCRIPTION:
This will be a randomized, single-blind, single-center, controlled, two arm, stratified (clinically diagnosed dentine hypersensitivity [DH] [Yes/No]), parallel group study to evaluate the efficacy of an experimental dentifrice containing 5% KNO3, 1% alumina and 5% STP, to maintain tooth color and reduce the accumulation of extrinsic tooth stain following peroxide tooth bleaching compared to a regular fluoride-containing dentifrice. The study will recruit generally healthy participants who wish to undergo peroxide tooth bleaching. Sufficient participants will be screened to randomize approximately 160 participants to study treatment to ensure approximately 128 evaluable participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is between the ages of 18-65 years, inclusive.
* Participant is willing and able to comply with scheduled visits, and other study procedures and restrictions.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history (for example, a medical condition confirmed to be causing xerostomia), or upon oral examination, that would impact the participant's safety, wellbeing or the outcomes of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Participant who is willing and able to undergo at-home tooth bleaching with peroxide containing treatment unsupervised.
* Participant with generally good oral health that fulfil all of the following:

  1. Teeth suitable for peroxide bleaching and gradable for tooth color and suitable for MLSI evaluation with no significant defects, calculus, restorations, crowns or veneers that could impact peroxide tooth bleaching performance or study evaluations as judged by the clinical examiner.
  2. Facial surfaces of maxillary anterior 6 teeth (tooth numbers 6-11) [Universal tooth number system] with mean Vita Bleached guide shade greater than or equal to (>=)13 at Visits 1 and 2.
  3. Having no lesions of the teeth or oral cavity that could interfere with the study evaluations.
  4. Having a minimum of 16 natural teeth.

Exclusion Criteria:

* Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 60 days prior to study entry and/or during study participation.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study or who is breastfeeding.
* Participant with known or suspected intolerance or hypersensitivity to the study materials [including the peroxide bleaching treatment] (or closely related compounds) or any of their stated ingredients.
* Participant who, in the opinion of the investigator or medically qualified designee, has a condition that would impact on their safety or wellbeing or affect their ability to understand and follow study procedures and requirements or who should not participate in the study for other reasons.
* Participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant with gross periodontal disease or who has had treatment for periodontal disease (including surgery) within 12 months of Screening or who has had scaling or root planning within 3 months of Screening.
* Participant who has had a peroxide tooth bleaching procedure (either professionally dispensed or at-home [including peroxide-containing dentifrices]) within 12 months of Screening.
* Participant who has had a dental prophylaxis within 8 weeks of screening.
* Participant who has used tooth desensitizing treatment (for example dentifrice, mouthwash et cetera) within 2 weeks of screening.
* Participant with a fixed or removable partial prosthesis, multiple dental implants or orthodontic braces/bands or fixed retainer or togue/lip piercing which, in the opinion of the investigator, could impact study outcomes.
* During the study period, participant taking daily doses of medication/treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of tooth sensitivity (examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquillizers, antidepressants, mood-altering and anti-inflammatory drugs). Participant will be allowed to use analgesics ad hoc to manage pain.
* Participant who has tooth abnormalities such as cracking or gross caries lesions that may, in the opinion of the investigator, impact the ability to evaluate tooth sensitivity.
* Participant who has previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 178 participants were screened into the study, 160 participants were enrolled and randomized to treatment (79 participants in the test dentifrice group and 81 participants in the reference dentifrice group). A total of 154 randomized participants completed the study.
Groups:
- Test Dentifrice: Participants dosed the toothbrush provided with a strip of test dentifrice (5 percent [%] Potassium nitrate [KNO3], 1% alumina, 5% Sodium tripolyphosphate [STP] and 1150 parts per million [ppm] fluoride as sodium fluoride) and brushed for two timed minutes twice daily (morning and evening) for up to 27 weeks (dentifrice was used for 2 weeks pre peroxide, 1 week during peroxide and 24 weeks post peroxide application). At Week 3, participants performed the first application of peroxide tooth bleaching as per the instructions provided and continued the application daily for up to 7 days.
- Reference Dentifrice: Participants dosed the toothbrush provided with a strip of reference dentifrice (dentifrice containing 1150 ppm fluoride as sodium fluoride) and brushed for two timed minutes twice daily (morning and evening) for up to 27 weeks (dentifrice was used for 2 weeks pre peroxide, 1 week during peroxide and 24 weeks post peroxide application). At Week 3, participants performed the first application of peroxide tooth bleaching as per the instructions provided and continued the application daily for up to 7 days.
Period: Overall Study
Arm/Group | Test Dentifrice | Reference Dentifrice
Started | 79 | 81
Completed | 75 | 79
Not Completed | 4 | 2
Not completed — Did not meet study criteria | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population comprised all randomized participants who received at least one dose of the study product.
Groups:
- Test Dentifrice: Participants dosed the toothbrush provided with a strip of test dentifrice (5% KNO3, 1% alumina, 5% STP and 1150 ppm fluoride as sodium fluoride) and brushed for two timed minutes twice daily (morning and evening) for up to 27 weeks (dentifrice was used for 2 weeks pre peroxide, 1 week during peroxide and 24 weeks post peroxide application). At Week 3, participants performed the first application of peroxide tooth bleaching as per the instructions provided and continued the application daily for up to 7 days.
- Total: Total of all reporting groups
Arm/Group | Test Dentifrice | Reference Dentifrice | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.91) | 37.6 (13.04) | 39.8 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 32 | 36 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 43
  Not Hispanic or Latino | 57 | 60 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 13 | 13 | 26
  Asian - East Asian Heritage | 1 | 1 | 2
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 4 | 6 | 10
  White - Arabic/North African Heritage | 4 | 3 | 7
  White - White/Caucasian/European Heritage | 42 | 41 | 83
  Multiple | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean VITA Shade Score at 24 Weeks After Tooth Bleaching
Description: Tooth color of the facial surfaces of the six anterior maxillary teeth was assessed by a single, trained clinical examiner using the VITA Bleachedguide 3D-MASTER. It consisted of a value-ranked ordered scale from 1 (the lightest) to 29 (the darkest). The shade level of each tooth surface was scored visually by the clinical examiner with reference to the Bleachedguide, where lower score indicated improvement.
Time Frame: At Week 24 after tooth bleaching
Population: The modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one assessment of tooth color after the bleaching period. Only those participants with data available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 75 | 79
score on a scale | 12.00 (0.355) | 12.06 (0.348)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Test type: Superiority; p = 0.9141, ANOVA; Adjusted Mean Difference = -0.05, 95% CI 2-sided [-1.04 to 0.93], Standard Error of Mean 0.498

2. Secondary Outcome: Adjusted Mean VITA Shade Score at 12 Weeks After Tooth Bleaching
Description: Tooth color of the facial surfaces of the six anterior maxillary teeth was assessed by a single, trained clinical examiner using the VITA Bleachedguide 3D-MASTER. It consisted of value-ranked ordered scale from 1 (the lightest) to 29 (the darkest). The shade level of each tooth surface was scored visually by the clinical examiner with reference to the Bleachedguide, where lower score indicated improvement.
Time Frame: At Week 12 after tooth bleaching
Population: The mITT population. Only those participants with data available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 72 | 77
score on a scale | 12.08 (0.353) | 11.71 (0.346)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Test type: Superiority; p = 0.4583, ANOVA; Adjusted Mean Difference = 0.37, 95% CI 2-sided [-0.61 to 1.34], Standard Error of Mean 0.494

3. Secondary Outcome: Adjusted Mean Total Modified Lobene Stain Index (MLSI) Score at 12 and 24 Weeks After Tooth Bleaching
Description: Extrinsic dental stain was assessed on the facial surfaces of the 6 maxillary anterior teeth using the MLSI. Area (A) and intensity (I) of extrinsic dental stain were scored separately for each tooth on the scale of 0 to 3 and the mean total score was presented, where 0=area with no stain, 1=Stain covering up to one third of area and light intensity stain, 2=Stain covering up to two thirds of area and moderate intensity stain, 3=Stain covering more than two thirds of area and heavy intensity stain. Total MLSI score = Area score multiplied by Intensity score and ranged from 0 to 9, where lower score indicated improvement.
Time Frame: At Week 12 and Week 24 after tooth bleaching
Population: The mITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 78 | 81
score on a scale
  Week 12: number analyzed (Participants) | 72 | 77
  Week 12 | 0.69 (0.044) | 0.87 (0.043)
  Week 24: number analyzed (Participants) | 75 | 79
  Week 24 | 0.72 (0.053) | 1.03 (0.052)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Week 12; Test type: Superiority; p = 0.0042, ANOVA; Adjusted Mean Difference = -0.18, 95% CI 2-sided [-0.30 to -0.06], Standard Error of Mean 0.061
Statistical Analysis 2: Comparison: Test Dentifrice vs Reference Dentifrice; Week 24; Test type: Superiority; p < 0.0001, ANOVA; Adjusted Mean Difference = -0.31, 95% CI 2-sided [-0.46 to -0.17], Standard Error of Mean 0.074

4. Secondary Outcome: Adjusted Mean MLSI Score at 12 and 24 Weeks After Tooth Bleaching in Gingival Sites, Interproximal Sites and Body Sites
Description: Extrinsic dental stain was assessed on the facial surfaces of the 6 maxillary anterior teeth using the MLSI. The facial surface of each assessable tooth was divided into individual sites. The gingival site was defined as a crescent-shaped band, approximately 2 millimeters wide, adjacent to the free margin of the gingiva and extending to the crest of the interdental papillae of the adjacent teeth. The remainder of the tooth surface was called as body site. Area (A) and intensity (I) of extrinsic dental stain were scored separately for each tooth on the scale of 0 to 3 and the mean score was presented, where 0=area with no stain, 1=Stain covering up to one third of area and light intensity stain, 2=Stain covering up to two thirds of area and moderate intensity stain, 3=Stain covering more than two thirds of area and heavy intensity stain. Total MLSI score = Area score multiplied by Intensity score and ranged from 0 to 9, where lower score indicated improvement.
Time Frame: At Week 12 and Week 24 after tooth bleaching
Population: The mITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 78 | 81
score on a scale
  Mean Gingival MLSI, Week 12: number analyzed (Participants) | 72 | 77
  Mean Gingival MLSI, Week 12 | 0.02 (0.012) | 0.03 (0.011)
  Mean Gingival MLSI, Week 24: number analyzed (Participants) | 75 | 79
  Mean Gingival MLSI, Week 24 | 0.01 (0.014) | 0.05 (0.014)
  Mean Interproximal MLSI, Week 12: number analyzed (Participants) | 71 | 77
  Mean Interproximal MLSI, Week 12 | 1.37 (0.088) | 1.71 (0.086)
  Mean Interproximal MLSI, Week 24: number analyzed (Participants) | 75 | 79
  Mean Interproximal MLSI, Week 24 | 1.44 (0.105) | 2.04 (0.103)
  Mean Body MLSI, Week 12: number analyzed (Participants) | 72 | 77
  Mean Body MLSI, Week 12 | 0.00 (0.007) | 0.01 (0.007)
  Mean Body MLSI, Week 24: number analyzed (Participants) | 75 | 79
  Mean Body MLSI, Week 24 | 0.00 (0.005) | 0.01 (0.004)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Gingival MLSI, Week 12; Test type: Superiority; p = 0.2478, ANOVA; Adjusted Mean Difference = -0.02, 95% CI 2-sided [-0.05 to 0.01], Standard Error of Mean 0.016
Statistical Analysis 2: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Gingival MLSI, Week 24; Test type: Superiority; p = 0.0957, ANOVA; Adjusted Mean Difference = -0.03, 95% CI 2-sided [-0.07 to 0.01], Standard Error of Mean 0.020
Statistical Analysis 3: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Interproximal MLSI, Week 12; Test type: Superiority; p = 0.0063, ANOVA; Adjusted Mean Difference = -0.34, 95% CI 2-sided [-0.58 to -0.10], Standard Error of Mean 0.122
Statistical Analysis 4: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Interproximal MLSI, Week 24; Test type: Superiority; p < 0.0001, ANOVA; Adjusted Mean Difference = -0.60, 95% CI 2-sided [-0.89 to -0.31], Standard Error of Mean 0.147
Statistical Analysis 5: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Body MLSI, Week 12; Test type: Superiority; p = 0.1536, ANOVA; Adjusted Mean Difference = -0.01, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.010
Statistical Analysis 6: Comparison: Test Dentifrice vs Reference Dentifrice; Mean Body MLSI, Week 24; Test type: Superiority; p = 0.1166, ANOVA; Adjusted Mean Difference = -0.01, 95% CI 2-sided [-0.02 to 0.00], Standard Error of Mean 0.006

5. Secondary Outcome: Adjusted Mean MLSI (Area) Score at 12 and 24 Weeks After Tooth Bleaching
Description: Extrinsic dental stain was assessed on the facial surfaces of the 6 maxillary anterior teeth using the MLSI. Area (A) of extrinsic dental stain was scored separately for each tooth on the scale of 0 to 3, where 0=area with no stain, 1=Stain covering up to one third of area, 2=Stain covering up to two thirds of area, 3=Stain covering more than two thirds of area. Total score ranged from 0 to 3, where lower score indicated improvement.
Time Frame: At Week 12 and Week 24 after tooth bleaching
Population: The mITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 78 | 81
score on a scale
  Week 12: number analyzed (Participants) | 72 | 77
  Week 12 | 0.55 (0.025) | 0.69 (0.024)
  Week 24: number analyzed (Participants) | 75 | 79
  Week 24 | 0.57 (0.027) | 0.74 (0.027)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Week 12; Test type: Superiority; p < 0.0001, ANOVA; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-0.21 to -0.07], Standard Error of Mean 0.035
Statistical Analysis 2: Comparison: Test Dentifrice vs Reference Dentifrice; Week 24; Test type: Superiority; p < 0.0001, ANOVA; Adjusted Mean Difference = -0.18, 95% CI 2-sided [-0.25 to -0.10], Standard Error of Mean 0.038

6. Secondary Outcome: Adjusted Mean MLSI (Intensity) Score at 12 and 24 Weeks After Tooth Bleaching
Description: Extrinsic dental stain was assessed on the facial surfaces of the 6 maxillary anterior teeth using the MLSI. Intensity (I) of extrinsic dental stain was scored separately for each tooth on the scale of 0 to 3, where 0=no stain, 1=light intensity stain, 2=moderate intensity stain, 3=heavy intensity stain. Total score ranged from 0 to 3, where lower score indicated improvement.
Time Frame: At Week 12 and Week 24 after tooth bleaching
Population: The mITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Dentifrice | Reference Dentifrice
Number analyzed (Participants) | 78 | 81
score on a scale
  Week 12: number analyzed (Participants) | 72 | 77
  Week 12 | 0.46 (0.023) | 0.52 (0.023)
  Week 24: number analyzed (Participants) | 75 | 79
  Week 24 | 0.48 (0.027) | 0.60 (0.026)
Statistical Analysis 1: Comparison: Test Dentifrice vs Reference Dentifrice; Week 12; Test type: Superiority; p = 0.0400, ANOVA; Adjusted Mean Difference = -0.07, 95% CI 2-sided [-0.13 to -0.00], Standard Error of Mean 0.033
Statistical Analysis 2: Comparison: Test Dentifrice vs Reference Dentifrice; Week 24; Test type: Superiority; p = 0.0010, ANOVA; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.20 to -0.05], Standard Error of Mean 0.037

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after the last administration of the study product or the last study procedure (up to approximately 195 days).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A serious adverse event (SAE) is a particular category of AE where the adverse outcome is serious.
Arm/Group | Test Dentifrice | Reference Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/79 | 1/81
Other Adverse Events (participants affected / at risk) | 39/79 | 42/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=79) | Reference Dentifrice (N=81)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Dentifrice (N=79) | Reference Dentifrice (N=81)
GINGIVAL PAIN (Gastrointestinal disorders) | 15 | 21
HYPERAESTHESIA TEETH (Gastrointestinal disorders) | 9 | 15
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 7 | 2
ANGULAR CHEILITIS (Gastrointestinal disorders) | 4 | 0
CHRONIC CHEEK BITING (Gastrointestinal disorders) | 3 | 1
GINGIVAL DISCOMFORT (Gastrointestinal disorders) | 3 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0
NONINFECTIVE GINGIVITIS (Gastrointestinal disorders) | 0 | 1
ORAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 15 | 19
GINGIVAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT06150573/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT06150573/SAP_001.pdf